CLINICAL TRIAL: NCT00615303
Title: The Effectiveness of Simethicone In Improving Visibility During Colonoscopy: A Randomized, Placebo-controlled Study
Brief Title: The Effectiveness of Simethicone In Improving Visibility During Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ramathibodi Hospital (Other)
Responsible Party: Principal Investigator, Abhasnee Sobhonslidsuk, Associate professor, Ramathibodi Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID12-49-23; ID12-49-23 (Other Grant/Funding Number: Gastroenterological Association of Thailand)
Record Dates: First submitted 2008-02-01; First posted 2008-02-14 (Estimated); Last update posted 2013-02-22 (Estimated); Status verified 2013-02

CONDITIONS: Colonoscopy
Keywords: Bowel preparation, colonoscopy, simethicone, air bubble
MeSH Terms: interventions — Simethicone; sodium phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 2 (Placebo Comparator)
  Interventions: Drug: Placebo
- 1 (Active Comparator)
  Interventions: Drug: Simethicone

INTERVENTIONS:
Drug: Simethicone — 2 dosages of either 45 ml of sodium phosphate plus 240 mg of simethicone tablets or 45 ml of sodium phosphate plus placebo in the evening before and in the morning of the procedure day. The colonoscopic examination was recorded
  Other Names: sodium phosphate
  Arms: 1
Drug: Placebo — 2 dosages of either 45 ml of sodium phosphate plus 240 mg of simethicone tablets or 45 ml of sodium phosphate plus placebo in the evening before and in the morning of the procedure day
  Other Names: Sodium phosphate
  Arms: 2

SUMMARY:
Sodium phosphate is one of the bowel preparation regimens for colonoscopy. However, intraluminal gas can impair visibility during the examination. Simethicone is medication that works by reducing the surface tension of air bubbles. We aimed to evaluate the effect of simethicone in enhancing visibility and efficacy during colonoscopy.

DETAILED DESCRIPTION:
A prospective, randomized, double-blinded, placebo-controlled study was conducted. One hundred and twenty-four patients were allocated to receive 2 dosages of either 45 ml of sodium phosphate plus 240 mg of simethicone tablets or 45 ml of sodium phosphate plus placebo in the evening before and in the morning of the procedure day. The colonoscopic examination was recorded. Visibility was blindly assessed for the amount of air bubbles and the degree of haziness by a single investigator. Five areas of the colon were graded for the amount of air bubbles, from 0 to 3; grade 0 and 1 were defined as the diminishing of air bubbles. The haziness was graded into 5 levels from excellent to unacceptable. Excellent, good and adequate were defined as the diminishing of haziness. The total duration of colonoscopy, the side effect of medication and the endoscopist and patient satisfaction were compared between 2 groups. Endoscopist satisfaction was evaluated by questionnaires. Visual analog scale (0-10) was used for rating patient satisfaction and the side effect of medication.

ELIGIBILITY:
Inclusion Criteria:

- Patients with age 18-70 yrs old who undergo colonoscopy at the endoscopic unit of the hospital

Exclusion Criteria:

* Renal insufficiency (Cr >2.3 mg/dl)
* Congestive heart failure
* Massive ascites
* Acute myocardial infarction within 6 months
* Coagulopathy
* Previous colonic surgery
* Suspected of colonic obstruction Pregnancy Refuse to give inform consent

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 194 (Actual)
Dates: Start 2006-12; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Visibility: air bubble and haziness | During colonoscopy

SECONDARY OUTCOMES:
Total colonoscopic time, patient and doctor satisfaction and side effects | During colonscopy

CONTACTS AND LOCATIONS:
Overall Officials: Abhasnee Sobhonslidsuk, M.D., Study Director — Ramathibodi Hospital
Locations (1):
- Ramathibodi hospital, Bangkok, Bangkok, Thailand